CLINICAL TRIAL: NCT06668753
Title: Effect of Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors on Non-alcoholic Fatty Liver Disease (NAFLD) in Type 2 Diabetic Patients with Diabetic Nephropathy
Brief Title: Effect of SGLT2 Inhibitors on NAFLD in Type 2 Diabetic Patients with Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Arafat Mahmoud Hassan, resident, Assiut University
Other Study IDs: Effect of SGLT2 I on NAFLD
Record Dates: First submitted 2024-09-06; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Effect of SGLT2 Inhibitors NAFLD in Type 2 Diabetic Patients with Diabetic Nephropathy
MeSH Terms: interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients: Dapagliflozin or Empagliflozin 10 mg once daily for 6 months
  Interventions: Drug: Dapagliflozin 10mg Tab or Empagliflozin 10 mg Tab
- controls: patients with standard anti-proteinuric regimen

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab or Empagliflozin 10 mg Tab — SGLT-2 inhibitors
  Groups: patients

SUMMARY:
To rule out the beneficial effect of SGLT2-I to reduce liver fat, and change in inflammatory markers (ALT, AST) in type 2 diabetic patients with non-alcoholic fatty liver disease.

And its role in improvement of Albuminuria and CKD progression.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD), is the most common liver disease and has been reported to be as high as 25%. It is characterized by the presence of fat in at least 5% of hepatocytes [1,2]. Lipid homeostasis in the liver is controlled by a very complex interplay between nuclear receptors, transcription factors, and hormones.

Excessive fat storage occurs when the balance between lipogenesis/lipid uptake versus lipid oxidation/excretion is disrupted [3,4]. NAFLD is usually associated with metabolic syndrome and is not, by definition, caused by excessive alcohol intake (defined as _20 g per day for women and _30 g per day for men) [1,2]. NAFLD represents a wide range of liver diseases, but histologically, it can be divided into two different types: non-alcoholic fatty liver (simple steatosis or NAFL) and non-alcoholic steatohepatitis (NASH), which is the more aggressive form [5-7]. Liver inflammation and injury are typical for NASH, and this form of NAFLD could lead to liver cirrhosis and hepatocellular cancer [2,8]. Due to the slow and asymptomatic progression of NAFLD, it is often diagnosed at a late stage. NAFLD has already become the second most common indication for liver transplantation. It takes around three to seven years for the development of NASH, which occurs in one-fifth of patients with NAFLD [9,10]. Currently, lifestyle modifications such as weight loss and physical activity are essential for all patients with NAFLD but are mostly not successful in the management of disease progression. Thus, there is an urgent need for approved medication therapy for NAFLD [4,5,11,12]. Ideal pharmacotherapy for NAFLD should decrease steatosis and inflammation, preferably liver fibrosis, while simultaneously improving insulin resistance, adiposity, and serum glucose levels [11]. There are currently numerous agents under clinical studies, and one of the leading candidates for Food and Drug Administration (FDA) approval is sodium-glucose cotransporter 2 (SGLT2) inhibitors [2,13,14]. Canagliflozin (Invokana), dapagliflozin, empagliflozin, ipragliflozin, tofogliflozin, and ertugliflozin, also known as "flozins", are glucose-lowering agents with an insulin-independent mode of action [15-19]. They were FDA-approved as oral antidiabetic drugs to reduce glucose levels by the inhibition of glucose reabsorption in the proximal renal tubule and are, in general, not associated with a risk of hypoglycaemia [20,21]. In general, SGLT2 inhibitors have a good safety profile, and the most frequent side effects reported are infection of the genitourinary tract and hypotension [16]. After gaining approval for T2DM, SGLT2 inhibitors were also approved for chronic kidney disease and heart failure in type 2 diabetic and the non-diabetic population due to their beneficial effects on the cardiovascular and renal systems [5,22]. In general, the antifibrotic and anti-inflammatory effects of SGLT2 inhibitors have been proposed as a common mode of action for liver, kidney, and heart protection [23]. Effect of SGLT2 Inhibitors on Liver is by conversion of carbohydrates from the bloodstream into fatty acids and ultimately into triglycerides or other lipids is a highly coordinated process called de novo lipogenesis [24]. Catabolism and lipolysis in extrahepatic tissues, especially adipose tissue, result in the transfer of free fatty acids to the liver, where excess fat results in liver steatosis. Insulin regulates both de novo lipogenesis and lipolysis. Since insulin resistance is usually present in NAFLD patients, insulin is unable to adequately inhibit adipose lipolysis [25]. Since insulin resistance is usually present in NAFLD patients, insulin is unable to adequately inhibit adipose lipolysis [25]. Furthermore, adipose tissue affects NAFLD progression by producing hormones and cytokines, which contribute to the dysfunction of hepatocytes and by increasing liver uptake of lipids [26]. Lipoprotein lipase (LPL), the enzyme that regulates the rate of hydrolysis of VLDL and triglycerides, is also involved in NAFLD development due to upregulation [4]. Dysregulation of liver lipid metabolism is associated with metabolic diseases such as T2DM and fatty liver. Regarding the pathophysiology of NAFLD improvement under SGLT-2i treatment, various mechanisms have been suggested. Treatment with SGLT-2i results in decreases in both glucose and insulin levels (especially in patients with DM), which lead to a large reduction of hepatic de novo lipid synthesis [27]. Moreover, glucagon-secreting alpha pancreatic cells also, express SGLT-2, thus the administration of SGLT-2i stimulates glucagon secretion [27,28,29]. In turn, the subsequently elevated plasma glucagon levels stimulate β- oxidation, and this shift from carbohydrate to fatty acid metabolism leads to reduced liver triglyceride content and consequently hepatic steatosis [27,30,31]. Another potential mechanism is mediated by the antioxidant effects of SGLT-2i. Apart from their ability to reduce high glucose-induced oxidative stress, SGLT-2i reduce free radical generation, suppress pro-oxidants, and upregulate antioxidant systems, such as superoxide dismutases (SODs) and glutathione (GSH) peroxidases [32,33,34,35,36,37].

ELIGIBILITY:
Inclusion Criteria:

-

Patients from 20 - 60 years old:

1. Patients Diagnosed as type 2 diabetes since ≥6 months
2. Patients Diagnosed with CKD GIII - IV non-HD
3. Patients Diagnosed with Metabolic associated fatty liver disease

Exclusion Criteria:

* 1. Type 1 diabetes or non-diabetic patients 2. BMI ≥40 kg/m2 3. Other causes of chronic liver disease (e.g., Hepatitis B virus, Hepatitis c virus, HIV, autoimmune disease, Wilson disease, drugs, alpha one antitrypsin deficiency).

  4. Patients use of drugs known to cause hepatic steatosis (e.g., amiodarone, valproate, tamoxifen, methotrexate, corticosteroids, contraceptive pills) 5. Detection of biliary duct obstruction based on imaging studies. 6. Patient with history of liver transplantation 7. liver cirrhosis (on basis of ultrasonography and MRI) or hepatocellular carcinoma (evidence on triphasic CT or MRI).

  8. Intolerance or allergy SGLT2-I or any other substance in the tablets. 9. Refused to consent to this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients presented to fibroscan clinic for evaluation of the degree of liver fibrosis and steatosis will be included in this study the data will be collected from Al-Rajhy hospital, Nephrology and Endocrinology units.
  About 114 patients all with basic antiproteinuric measures divided into two groups:
  A) Group 1(exposed): 57 patients given SGLT-2 inhibitors B) Group 2(non-exposed): 57 controls with no SGLT-2 inhibitors
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
effect of SGLT2-I on NAFLD | baseline
  To rule out the beneficial effect of SGLT2-I in changing liver fat using the fibroscan, and in changing hepatic inflammatory markers (ALT (SGPT) ranges from about 7-56 units/liter of serum, normal levels of AST (SGOT) is about 5-40 units/liter of serum) in type 2 diabetic patients with non alcoholic fatty liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Hussien Ahmed Elamin, PHD, Principal Investigator — Assiut University; Essam Abdel Aziz, PHD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No